CLINICAL TRIAL: NCT01121523
Title: Effect of Cue-based Tactile Stimulation on Premature, Low Birth Weight Infants: Stress Reactivity.Immune Functioning, and Parenting
Brief Title: Cue-based Tactile Stimulation and Infant Stress Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Douglas M. Teti, Professor of Human Development, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Project Touch
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Premature; Infant, Light-for-dates
Keywords: Prematurity; massage; stress; parenting; infancy; sleep; intervention
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cue-directed tactile stimulation (Experimental)
  Interventions: Behavioral: Cue directed tactile stimulation
- Control group (Active Comparator)
  Interventions: Behavioral: Cue directed tactile stimulation

INTERVENTIONS:
Behavioral: Cue directed tactile stimulation — Cue-based tactile stimulation delivered to medically stable premature infants three times daily by mothers or trained NICU nurses daily for 4 consecutive weeks
  Other Names: Massage

SUMMARY:
The present study is an examination of cue-directed tactile stimulation (CTDS), administered by mothers and NICU nurses, on infant and maternal stress reactivity, infant immune system functioning, maternal parenting cognitions, and parenting competence.

DETAILED DESCRIPTION:
The overarching aim of this study is to assess the effects of a program of mother-delivered, cue-based infant massage on stress reactivity in the mother-infant dyad, and on other measures of mother-infant functioning. The study has several interrelated objectives:

1. To evaluate the short-term effects of infant massage intervention on infant and maternal stress reactivity from assays of maternal and infant salivary cortisol, and cortisol levels in mothers' breast milk.
2. To examine the impact of mother-delivered infant massage on the development of infant resistance to infectious pathogens and antibody-based protective immunity in response to routine scheduled vaccinations, and to examine if the degree of immunity is mediated by infant stress reactivity.
3. To examine the impact of mother-delivered infant massage, and of changes in stress reactivity in response to massage, on infant physiological functioning (vagal tone, heart rate variability), infant physical development (weight, height, and head circumference), mothers' perception of infant temperament and infant state regulation, parenting self-efficacy, symptoms of depression and anxiety, and mother-infant interaction.
4. To examine associations between cortisol levels in mothers' saliva, mothers' breast milk, and infants' saliva. Establishing such linkages would support recent animal data suggesting that infant glucocorticoid levels can be affected by glucocorticoid levels transferred to the infant in mother's milk.
5. To examine whether a single nucleotide polymorphism (SNP) in three candidate genes (Mu opioid receptor, brain-derived neurotropic factor, and vasopressin V1b receptor), each associated with hypothalamic-pituitary-adrenal axis (HPA) functioning, moderates the effects of infant massage on stress-related outcomes.

ELIGIBILITY:
Exclusion Criteria:

* The following babies will be excluded:

  * With any chromosomal abnormality
  * With congenital heart disease
  * With any surgical intervention
  * With intraventricular hemorrhages greater than grade II
  * If mother dies during delivery

Ages: 7 Days to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Stress reactivity | one month post-intervention
  Infant and maternal salivary cortisol

SECONDARY OUTCOMES:
Infant immune functioning | 2-3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Douglas M Teti, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- Penn State Hershey Children's Hospital, Hershey, Pennsylvania, United States